CLINICAL TRIAL: NCT05777460
Title: Results From a Multicenter Registry on the Outcomes of the Terumo Custom-made Aortic Endograft
Brief Title: Mid- and Long-term Outcomes of Custom-made Aortic Devices
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2992
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Aortic Diseases; Thoracic Aortic Aneurysm
MeSH Terms: conditions — Aortic Diseases; Aortic Aneurysm, Thoracic | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Thoracic endovascular aortic repair (TEVAR) — The TEVAR procedure involves the placement of a covered stent (a metal mesh tube with a layer of fabric) into the weakened area of the artery.

SUMMARY:
This study aims to evaluate mid- and long-term outcomes after Thoracic endovascular aortic repair (TEVAR) with custom-made devices.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic Aortic Disease

Exclusion Criteria:

* Urgent/Emergent treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients that underwent Thoracic Endovascular Aortic Repair (TEVAR) in the period 2015-2023 with the Custom Relay® Multi-Feature™ Terumo Aortic will be included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall Mortality | 3 years
  Any death occurring during follow-up
Aortic-related mortality | 3 years
  Any death occurring during follow-up and related to the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No